CLINICAL TRIAL: NCT02387801
Title: Early Onset of Clinical Improvement With Ixekizumab in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of the Early Activity of Ixekizumab (LY2439821) in Moderate-to-Severe Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15454; I1F-US-RHBO (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ixekizumab Dosing Q2W (Experimental): 160 milligrams (mg) ixekizumab given as two subcutaneous (SC) injections at week 0 followed by 80 mg ixekizumab given as a single SC injection once (Q2W) every 2 weeks through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 44.
  Interventions: Drug: Ixekizumab
- Ixekizumab Dosing Q4W (Experimental): 160 mg ixekizumab given as two SC injections at week 0 followed by 80 mg ixekizumab given as a single SC injection once (Q4W) every 4 weeks through week 44.
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821

SUMMARY:
To detect onset of activity of ixekizumab in participants with moderate-to-severe plaque psoriasis and to document the same using sequential photographic images.

ELIGIBILITY:
Inclusion Criteria:

* Present with chronic moderate-to-severe plaque psoriasis based on a confirmed (by a dermatologist) diagnosis of chronic plaque psoriasis for at least 6 months prior to baseline
* Active psoriatic skin lesions of plaque psoriasis (Ps)
* Are a candidate for phototherapy and/or systemic therapy
* Men must agree to use a reliable method of birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment
* Women must agree to use reliable birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment

Exclusion Criteria:

* Are unable to commit to the photography schedule for the duration of the study
* Have participated in any study with interleukin 17 (IL-17) or (IL-23) antagonists, including ixekizumab
* Serious disorder or illness other than psoriasis
* Serious infection within the last 3 months
* Breastfeeding or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Mount Sinai School of Medicine Dermatology Clinical Trials, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Background] Khattri S, Goldblum O, Solotkin K, Amir Y, Min MS, Ridenour T, Yang FE, Lebwohl M. Early Onset of Clinical Improvement with Ixekizumab in a Randomized, Open-label Study of Patients with Moderate-to-severe Plaque Psoriasis. J Clin Aesthet Dermatol. 2018 May;11(5):33-37. Epub 2018 May 1. PMID 29785237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Induction Dosing Period (Weeks 0 up to 12), Maintenance Dosing Period (Weeks 12 up to 48), Minimum Post Treatment Follow-Up Period up to 12 weeks after last visit.
Pre-assignment Details: Participants were randomized to ixekizumab (ixe) 80 mg Q2W or Q4W during the Induction Dosing Period from Week 0 to Week 12. Participants received ixe Q4W in the Maintenance Dosing Period from Week 12 to Week 48, and then to the Post Follow up Treatment Period for at least 12 weeks.
Groups:
- Ixekizumab Q2W: 160 milligrams (mg) ixekizumab given as two subcutaneous (SC) injections at week 0 followed by 80 mg ixekizumab given as a single SC injection once (Q2W) every 2 weeks through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 44.
- Ixekizumab Q4W: 160 mg ixekizumab given as two SC injections at week 0 followed by 80 mg ixekizumab given as a single SC injection once (Q4W) every 4 weeks through week 44.
Period: Induction Dosing Period
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Maintenance Dosing Period
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W
Started | 0 (All participants from Induction Dosing Period went to ixe Q4W arm during Maintenance Dosing Period.) | 12
Completed | 0 | 12
Not Completed | 0 | 0
Period: Post-Treatment Follow-up
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W
Started | 0 | 12
Completed | 0 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ixekizumab Q2W: 160 mg ixekizumab given as two SC injections at week 0 followed by 80 mg ixekizumab given as a single SC injection once Q2W through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 44.
- Ixekizumab Q4W: 160 mg ixekizumab given as two SC injections at week 0 followed by 80 mg ixekizumab given as a single SC injection once Q4W through week 44.
- Total: Total of all reporting groups
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (12.54) | 55.2 (7.39) | 48.5 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to at Least a 1 Point Improvement on the Patient's Global Assessment of Disease Severity (PatGA) Score
Description: The PatGA is a patient-administered single-item scale on which participants are asked to rank by selecting a number on a 0 to 5 Numeric Rating Score (NRS) the severity of their psoriasis "today" from 0 (Clear) = no psoriasis to 5 (Severe) = the worst their psoriasis has ever been.
Time Frame: Baseline through Week 12
Population: All randomized participants.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W
Number analyzed (Participants) | 6 | 6
Days | 5.0 [2.0 to 5.0] | 6.0 [4.0 to 7.0]

2. Secondary Outcome: Mean Change From Baseline on Itch Numeric Rating Scale (NRS) Score
Description: The Itch NRS is a patient-administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching from psoriasis (Ps) is indicated by circling the number that best describes the worst level of itching in the past 24 hours. Least Square Means (LS means) are from analysis of mixed-effects model for repeated measures (MMRM) and model includes treatment group, baseline value and timepoint.
Time Frame: Baseline, Week 12
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W
Number analyzed (Participants) | 6 | 6
units on a scale | -6.2 (0.53) | -6.6 (0.55)

3. Secondary Outcome: Mean Change From Baseline on the Dermatology Life Quality Index (DLQI)
Description: The DLQI is a simple, patient-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". For all questions, if unanswered the question is scored as "0". Totals range from 0 to 30 (less to more impairment). LS means are from analysis of MMRM and model includes treatment group, baseline value and timepoint.
Time Frame: Baseline, Week 12
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W
Number analyzed (Participants) | 6 | 6
units on a scale | -13.4 (1.56) | -14.3 (1.59)

4. Secondary Outcome: Mean Change From Baseline in Percent Body Surface Area (%BSA)
Description: The BSA is the percentage involvement of psoriasis on each participant's body surface on a continuous scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participant's hand (including the palm, fingers, and thumb). The total BSA affected was the summation of individual regions affected. LS means are from analysis of MMRM and the model includes treatment group, baseline value, visit and treatment-by-visit interaction
Time Frame: Baseline, Week 12
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W
Number analyzed (Participants) | 6 | 6
percentage of body surface area | -26.1 (1.39) | -28.0 (1.39)

5. Secondary Outcome: Mean Change From Baseline on the Psoriasis Area and Severity Index (PASI)
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 75 were defined as having an improvement of at least 75% in PASI scores compared to baseline. LS means are from analysis of MMRM and the model includes treatment group, baseline value, visit and treatment-by-visit interaction.
Time Frame: Baseline, Week 12
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W
Number analyzed (Participants) | 6 | 6
units on a scale | -22.00 (0.456) | -22.72 (0.456)

6. Secondary Outcome: Time to at Least a 2 Point Improvement on the PatGA Score
Description: The PatGA is a patient-administered single-item scale on which participants are asked to rank by selecting a number on a 0 to 5 NRS the severity of their psoriasis "today" from 0 (Clear) = no psoriasis to 5 (Severe) = the worst their psoriasis has ever been.
Time Frame: Baseline though Week 12
Population: All randomized participants.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Ixekizumab Q2W | Ixekizumab Q4W
Number analyzed (Participants) | 6 | 6
Days | 10.0 [6.0 to 12.0] | 13.5 [5.0 to 22.0]

ADVERSE EVENTS:
Groups:
- Ixekizumab Q2W Induction Dosing Period: 160 mg ixekizumab given as two SC injections at week 0 followed by 80 mg ixekizumab given as a single SC injection once Q2W through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 44.
- Ixekizumab Q4W Induction Dosing Period: 160 mg ixekizumab given as two SC injections at week 0 followed by 80 mg ixekizumab given as a single SC injection once Q4W through week 44.
- Ixekizumab 80 mg Q4W Maintenance: After week 12 all participants are given 80 mg ixekizumab as a single SC injection once Q4W through week 44.
- Ixekizumab 80 mg Q4W Post-treatment: All participants receiving at least one dose of ixekizumab entered the post treatment follow-up period for a minimum of 12 weeks.
Arm/Group | Ixekizumab Q2W Induction Dosing Period | Ixekizumab Q4W Induction Dosing Period | Ixekizumab 80 mg Q4W Maintenance | Ixekizumab 80 mg Q4W Post-treatment
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6 | 9/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab Q2W Induction Dosing Period (N=6) | Ixekizumab Q4W Induction Dosing Period (N=6) | Ixekizumab 80 mg Q4W Maintenance (N=12) | Ixekizumab 80 mg Q4W Post-treatment (N=12)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Biopsy breast (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Biopsy prostate (Investigations) | 0/5 (0) | 1/3 (1) | 0/8 (0) | 0/8 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye laser surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days